CLINICAL TRIAL: NCT07192653
Title: Intraoperative Endovascular Treatment Via the Ligamentum Teres Hepatis in Liver Transplantation for Yerdel Grade Ⅲ/IV Portal Vein Thrombosis: A Safe and Effective Strategy
Status: Completed | Type: Observational
Sponsor: Chiyi Chen (Other)
Responsible Party: Sponsor-Investigator, Chiyi Chen, Attending physician, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Other Study IDs: ChenC
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplantation; Endovascular Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Period 1
  Interventions: Procedure: nonanatomical anastomosis
- Period 2
  Interventions: Procedure: LTH-based EVT

INTERVENTIONS:
Procedure: nonanatomical anastomosis — In Period 1 (2016-2019, n=41), nonanatomical anastomosis was performed if portal flow was insufficient.
  Groups: Period 1
Procedure: LTH-based EVT — In Period 2 (2019-2024, n=34), patients with persistent hypoperfusion underwent additional LTH-based EVT (stenting or shunt occlusion)
  Groups: Period 2

SUMMARY:
Background: To evaluate the safety and efficacy of intraoperative endovascular treatment (EVT) using the donor ligamentum teres hepatis (LTH) approach for Yerdel grade III/IV portal vein thrombosis (PVT) during liver transplantation (LT), a condition that poses a major challenge in complex surgeries.

Methods: This single-center retrospective cohort study included some patients with grade III/IV PVT who underwent LT and were divided into two periods: in both periods, patients underwent modified eversion thrombectomy. However, in Period 1 (2016-2019), nonanatomical anastomosis was performed if portal flow was insufficient, and in Period 2 (2019-2024), patients with persistent hypoperfusion underwent additional LTH-based EVT (stenting or shunt occlusion). Perioperative outcomes (operative time, anhepatic phase, and anastomosis type) and long-term outcomes (graft survival and complication rates) were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years).
* Patients underwent deceased-donor liver transplantation.
* At Tianjin First Central Hospital between February 2016 and December 2024.
* Identified recipients with Yerdel grade III/IV PVT, which was confirmed by multiphase contrast-enhanced CT, indirect portography, and intraoperative evaluation

Exclusion Criteria:

* Exclusion criteria were living-donor and split-liver procedures.
* All procedures were performed using classic orthotopic transplantations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Conducted a retrospective cohort analysis of 1,478 consecutive adult patients (aged ≥18 years) who underwent deceased-donor liver transplantation at Tianjin First Central Hospital between February 2016 and December 2024.From this population, the investigators identified 75 recipients with Yerdel grade III/IV PVT, which was confirmed by multiphase contrast-enhanced CT, indirect portography, and intraoperative evaluation. Exclusion criteria were living-donor and split-liver procedures. All procedures were performed using classic orthotopic transplantations. To evaluate the evolution of our PVT management strategy, the investigators divided the cohort into two chronologically distinct periods: period 1 (pre-intervention): February 2016-January 2019 (n=41), and period 2 (LTH protocol): February 2019-December 2024 (n=34).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-04 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intraoperative
  Operative time refers to the duration from the initial surgical incision to the completion of skin closure.
Anhepatic Phase Time | Intraoperative
  The anhepatic phase time is the critical period during liver transplant surgery when the patient's native liver has been removed and the donor liver has not yet been reperfused.
Rate of Nonanatomical Reconstruction | Intraoperative
  The rate of nonanatomical resection refers to the frequency with which a surgical procedure removes a tumor without following the boundaries of the organ's functional anatomical units.
Delayed Graft Function | Within 7 days postoperatively
  Delayed graft function is a common complication following kidney transplantation where the transplanted organ does not function immediately, often necessitating dialysis within the first week post-surgery.
Portal Vein Complications | From the surgery to the last follow-up (median follow-up 28 months)
  Portal vein complications are a serious concern in liver transplantation, encompassing issues such as thrombosis, stenosis, and occlusion that can threaten graft survival and patient life.
Graft Survival | 1-year and 3-year postoperatively
  Graft survival refers to the continued functional existence of a transplanted organ or tissue within a recipient's body.

IPD SHARING:
Plan to Share IPD: No